CLINICAL TRIAL: NCT06802796
Title: Plasma NGAL as a Predictor to Acute Pyelonephritis : Case -Control Cohort Study .
Brief Title: Plasma NGAL in APN Patients
Status: Completed | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelhalim Elsayed, assistant lecturer of urology, Kafrelsheikh University
Other Study IDs: KFSIRB200-143
Record Dates: First submitted 2025-01-25; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pyelonephritis
MeSH Terms: conditions — Pyelonephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A :patient with pyelonephritis: patient with pyelonephritis
  Interventions: Diagnostic Test: Plasma NGAL test
- Group B :patient without pyelonephritis: patient without pyelonephritis
  Interventions: Diagnostic Test: Plasma NGAL test

INTERVENTIONS:
Diagnostic Test: Plasma NGAL test — Human neutrophil gelatinase-associated lipocalin ELISA Kit from BT LAB® Bioassay technology laboratory was used for the estimation of serum NGAL. Procedure was done according to the manufacturer's instructions.

SUMMARY:
In recent years, novel biomarkers of renal dysfunction have attracted attention for the diagnosis of UTIs. NGAL is a 25 kDa protein that belongs to the lipocalin. It acts as a transporter for small hydrophobic molecules and is involved in many physiological processes, such as modulating inflammation, innate immune response, and maintaining metabolic homeostasis

ELIGIBILITY:
Inclusion Criteria:

* above 20 years Suspected have pyelonphirtis

Exclusion Criteria:

* age below 20

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patient had fever due to renal infection
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Result of plasma NGAL test | One day
  Result of serum test of NGAL

CONTACTS AND LOCATIONS:
Locations (1):
- Elsayed Abdelhalim Elsayed, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided